CLINICAL TRIAL: NCT00738738
Title: A Phase 3, 6-Month Open-Label Safety Study Of PD 0332334 In Elderly Patients With Generalized Anxiety Disorder
Brief Title: 6-Month Open-Label Safety Study Of PD 0332334 In Elderly Patients With Generalized Anxiety Disorder (GAD)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Please see Detailed Description for termination reason.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5361036
Record Dates: First submitted 2008-08-12; First posted 2008-08-20 (Estimated); Last update posted 2012-12-03 (Estimated); Status verified 2012-11

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder Elderly
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — imagabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: PD-0332334 — Dosage from: 50-100 mg oral capsule Dosage and frequency: 50-350 mg once or twice a day Duration: 6 months
  Other Names: imagabalin

SUMMARY:
This is an open-label, multi-site, 6-month study of an investigational compound in elderly outpatients, age 65 years old or above, to assess the long-term safety and tolerability of the compound in the treatment of elderly subjects with Generalized Anxiety Disorder (GAD).

DETAILED DESCRIPTION:
Termination reason: On February 23rd 2009, a decision to terminate further development for PD 0332334 was communicated to investigators in this study. The decision to terminate this study was not based on any safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age > 65 years.
* A primary diagnosis of Generalized Anxiety Disorder according to the Diagnostic and Statistical Manual-IV (DSM-IV).
* Subjects must have a HAM-A score of 16 or higher at both screening and baseline visits.

Exclusion Criteria:

* Women who are pregnant or contemplating pregnancy (eg, via in vitro fertilization) during the study through 30 days after the last dose of study medication.
* Subjects with evidence of a current (within the past 6 months) clinically significant or unstable hematological, autoimmune, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, pancreatic, psychiatric, neurologic, immunological or retinal disorder; subjects with an active infection within the past 2 months.
* Subjects who have an ongoing, unresolved, clinically significant cardiovascular or cerebrovascular medical problem.
* Mini Mental Status Exam (MMSE) score <24 or possibility of undiagnosed dementia, cognitive or amnestic disorder, including, but not limited to mild cognitive impairment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Discontinuations due to adverse events or adverse events occurring during and after the discontinuation of trial medication | Weekly
The nature, incidence, duration, and severity of adverse events. | Weekly
Suicide related adverse events will be further assessed using the Columbia Suicide Severity Rating Scale as needed | As needed
The primary outcome is safety which will be assessed throughout the 6-months by physical exams, monitoring of vital signs, body weight changes, and clinical safety laboratory | Screening, Baseline, Wk 4, Wk 14, Wk 26/EOT, & at FU; Vital signs at every vist
Electrocardiograms will be performed to assess any changes in cardiac functioning related to the compound | Screening, Baseline, Wk 4, Wk 15 & Wk 26/EOT

SECONDARY OUTCOMES:
Symptom severity of generalized Anxiety Disorder (GAD) will be measured by the Hamilton Rating Scale for Anxiety (HAM-A). | Screening, Baseline, Wk 1-2, Wk 4, Wk 14, Wk 26/EOT & Wk 27 (FU)
Overall Health Care utilization will be assessed with the Health Care Utilization (HCU) questionnaire. | Twice at Wk 13 and Wk 26/EOT
Also, the Daily Diary (including the Daily assessment of Symptoms DAS-A and Global Anxiety - Visual Analog Scale (GA-VAS) and the Clinical Global Impression of Severity (CGI-S) will be used to assess symptoms of GAD. | Screening, Baseline, Wk 1-2, Wk 4, Wk 14, Wk 26/EOT
Plasma concentrations will be collected to evaluate the population pharmacokinetics and the dose/exposure relationships for safety and efficacy . | 1 time

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Prairie Village, Kansas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5361036&StudyName=6-Month%20Open-Label%20Safety%20Study%20Of%20PD%200332334%20In%20Elderly%20Patients%20With%20Generalized%20Anxiety%20Disorder%20%28GAD%29